CLINICAL TRIAL: NCT01036321
Title: Phase II Clinical Trial of Purified Isoflavones in Prostate Cancer: Comparing Safety, Effectiveness and Mechanism of Action Between African American and Caucasian Men
Brief Title: Phase II Clinical Trial of Purified Isoflavones in Prostate Cancer: Comparing Safety, Effectiveness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCC-15835; IRB 107980 (Other: USF IRB); 1P20MD003375-01 (NIH)
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Purified Isoflavones (Active Comparator): Soy-based isoflavone concentrate with methyl cellulose blend filler. 40 mg daily.
  Interventions: Drug: Purified isoflavones
- Methyl cellulose blend (Placebo Comparator): Placebo.
  Interventions: Drug: Methyl cellulose blend

INTERVENTIONS:
Drug: Purified isoflavones — Soy-based isoflavone concentrate with methyl cellulose blend filler - Take 2 capsules daily
  Other Names: Novasoy 400; Avicel PH105
  Arms: Purified Isoflavones
Drug: Methyl cellulose blend — Placebo - Take 2 capsules daily
  Other Names: Avicel PH105
  Arms: Methyl cellulose blend

SUMMARY:
The purpose of our study is to recruit and treat 96 men diagnosed with prostate cancer and scheduled for a prostatectomy with a capsule form of either purified isoflavones or placebo for a 3-6 week period to see if we can slow down the rate of prostate cancer growth. A placebo is a pill or something that looks like the medicine that is being studied but has no active medicine in it. We also want to see if taking purified isoflavones is safe and if it reduces lower urinary tract symptoms. In addition, we want to study if purified isoflavones are able to slow the progression of prostate cancer, and the mechanism of action of purified isoflavones. If the safety and the effects of purified isoflavones on slowing down the progression of prostate cancer is shown in our study, this will also be a safe way of treating men who are at high risk of prostate cancer, so that we can prevent prostate cancer in the future.

DETAILED DESCRIPTION:
Patients will need to take two (2) capsules daily, one with their breakfast and one with their dinner. On the day prior or the day that patients are coming in for their pre-operative surgery blood work, we ask that they take the second dose with lunch, if their appointment is in the afternoon.

At the start of the study and at the end of the study (3-6 weeks), patients will undergo interviews, complete questionnaires, and have lab tests to determine if this drug is effective to reduce progression of prostate cancer and is safe to use.

Patients will also receive a multivitamin/mineral supplement for the 3-6 weeks that they are on this study and will be required to take one (1) every day. It is required that patients not take any other vitamin/mineral or herbal preparation containing isoflavones and avoid eating or drinking soy products.

We anticipate that most patients will be scheduled for a prostatectomy 3-6 weeks (+/- 3 days) from start of study agent. In addition to their first visit, patients will be required to come in the day of the surgery for prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of localized prostate cancer (PCa), based on pathological assessment from biopsy specimens
* No prior or current therapy for PCa or history of cancer except non-melanoma skin cancer
* Scheduled for prostatectomy between 3- 6 weeks (+/-3 days) after start of study agent
* No known history of hepatic or renal disease (LFTs (SGOT/SGPT) > 5.0 x upper limit of normal as evidenced by impairment of baseline laboratory values, Actual creatinine clearance of >60 utilizing the Cockcroft-Gault formula (1976), which employs creatinine measurements and a patient's weight to predict the clearance. The constant is 1.23 for men.
* Omnivorous diet
* No evidence of prostatitis or urinary tract infection
* Able and willing to give written informed consent
* Currently not using or willing to discontinue any nutritional supplements that contain soy or soy isoflavones
* Not allergic to study supplements
* Not on antibiotics
* Men who do not consume more than 3 - 4 oz. of soy or soy products per week
* Not taking steroid hormones or medications which have known impact on prostatic specific antigen (PSA)
* Health status cleared by primary MD or urologist
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Exclusion Criteria:

* Prior history of prostate cancer; Current or prior history of other malignancies (exceptions include nonmelanoma skin cancer or other cancer with no evidence of tumor recurrence five years after definitive treatment)
* History of renal or hepatic disease, including history of hepatitis B, C or delta as evidenced by impairment of baseline laboratory values
* Participation in any other investigational study or use of any other investigational agents within 30 days of study entry
* History of allergic reactions attributed to soy isoflavones or other compounds of similar chemical or biologic composition to Novasoy 400® or the inactive components present in the purified isoflavone and placebo capsules
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any psychological, familial, sociological or other concomitant condition that would not allow adequate compliance with the study protocol
* Only African American (a person having origins in any of the black racial groups of Africa) and Caucasian (a person having origins in any of the original people of Europe, Middle East, or North Africa) men, as defined by the NIH, will be included in this study. Since this is an investigation targeting men with PCa, women are not eligible for the study.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-12-11 (Actual); Primary Completion 2014-06-26 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - University of Florida & Shands Medical Center - Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - James A. Haley VA Hospital, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from January 2010 through May 2014 at three sites in Florida.
Pre-assignment Details: 75 were consented and were further screened for final eligibility. 3 were ineligible and 1 withdrew after screening, before randomization. 71 were randomized. 1 was ineligible after randomization.
Groups:
- Active Comparator: Purified Isoflavones: Soy-based isoflavone concentrate with methyl cellulose blend filler - 2 capsules daily.
- Placebo Comparator: Methyl Cellulose Blend: Placebo: Methyl cellulose blend - 2 capsules daily.
Period: Overall Study
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Started | 36 | 35
Completed | 31 | 31
Not Completed | 5 | 4
Not completed — Ineligible after randomization | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to a study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (7.5) | 59.1 (7.4) | 58.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 35 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 28 | 25 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Percent Ki-67 From Baseline
Description: Efficacy: Change in percent Ki-67 evaluated in prostate cancer (PCa) tissue specimens after 3-6 weeks of intervention with purified isoflavones (40 mg daily) vs. Placebo.
Time Frame: Baseline to post intervention - up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: percentage of tumor cells
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
percentage of tumor cells
  All Participants | 0.5 [0.0 to 2.0] | 1.0 [0.0 to 6.0]
  Caucasian Men (CM) | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 6.0]
  African American Men (AAM) | 0.3 [0.0 to 0.5] | 1.0 [1.0 to 1.0]

2. Primary Outcome: Number of Toxicity Events by Final Attribution and Treatment Arm
Description: Safety: Incidence of Adverse Events (AEs) occurring during intervention with either 20 mg purified isoflavones bid or placebo. Serious Adverse Event (SAEs) and other Adverse Event (AE) details are also reported in the Adverse Event sections.
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Number; unit: Toxicity Events
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
Toxicity Events
  Possibly related | 37 | 37
  Probably related | 4 | 0
  Relation unlikely | 17 | 9
  Unrelated | 24 | 20
  Total | 82 | 66

3. Secondary Outcome: Biomarkers of Disease Progression - Serum PSA
Description: Median change from baseline to post intervention: Prostatic specific antigen (PSA). All Participants (ALL); Caucasian Men only (CM only); African American Men only (AAM only).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
ng/mL
  ALL | -0.7 [-3.5 to 1.2] | -0.2 [-3.2 to 2.7]
  CM only | -0.8 [-3.5 to 1.2] | -0.2 [-2.9 to 2.7]
  AAM only | -0.3 [-2.5 to 1.2] | -1.0 [-3.2 to 2.0]

4. Secondary Outcome: Change in Plasma Concentrations of Isoflavone
Description: Plasma concentrations of isoflavone: Genistein from baseline to post intervention by study arm.
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: mg
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
mg | 0.00 [-3.06 to 0.37] | -0.02 [-1.36 to 0.47]

5. Secondary Outcome: Biomarkers of Disease Progression - Estradiol
Description: Median change from baseline to post intervention. Steroid hormones: pre-treatment (Pre:) versus post treatment (Post:).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: pmo/L
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
pmo/L
  Pre: Estradiol pmo/L | 37.5 [18.0 to 67.0] | 37.0 [17.0 to 67.0]
  Post: | 39.0 [15.0 to 71.0] | 39.5 [17.0 to 60.0]

6. Secondary Outcome: Biomarkers of Disease Progression - Free Testosterone
Description: Median change from baseline to post intervention. Steroid hormones: pre-treatment (Pre:) versus post treatment (Post:).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
pg/ml
  Pre: Free testosterone (pg/ml) | 59.9 [21.3 to 101.0] | 49.1 [30.4 to 134.0]
  Post: | 54.8 [17.6 to 119.0] | 62.9 [24.8 to 106.0]

7. Secondary Outcome: Biomarkers of Disease Progression - Insulin Like Growth Factor (IGF) Binding Protein -3
Description: Median change from baseline to post intervention. Steroid hormones: pre-treatment (Pre:) versus post treatment (Post:).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
mg/L
  Pre: IGF Binding Protein -3 (mg/L) | 3.9 [1.8 to 5.5] | 4.3 [1.7 to 6.4]
  Post: | 3.8 [1.7 to 4.7] | 4.2 [2.0 to 5.6]

8. Secondary Outcome: Biomarkers of Disease Progression - IGF-1
Description: Median change from baseline to post intervention. Steroid hormones: pre-treatment (Pre:) versus post treatment (Post:).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
ng/mL
  Pre: IGF-1 (ng/mL) | 160.0 [0.0 to 288.0] | 143.0 [52.0 to 285.0]
  Post: | 153.0 [53.0 to 258.0] | 143 [71.0 to 301.0]

9. Secondary Outcome: Biomarkers of Disease Progression - Sex Hormone-binding Globulin (SHBG)
Description: Median change from baseline to post intervention. Steroid hormones: pre-treatment (Pre:) versus post treatment (Post:).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: nmol/L
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
nmol/L
  Pre: SHBG nmol/L | 34.0 [14.0 to 92.0] | 32.0 [12.0 to 110.0]
  Post: | 35.0 [13.0 to 61.0] | 32.0 [14.0 to 81.0]

10. Secondary Outcome: Biomarkers of Disease Progression - Total Testosterone
Description: Median change from baseline to post intervention. Steroid hormones: pre-treatment (Pre:) versus post treatment (Post:).
Time Frame: Up to 6 weeks
Population: All participants who were randomized to a study arm.
Measure: Median (Full Range); unit: ng/dL
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Number analyzed (Participants) | 36 | 35
ng/dL
  Pre: Total Testosterone (ng/dL) | 358.0 [93.0 to 738.0] | 348.0 [179.0 to 979.0]
  Post: | 376.0 [163.0 to 709.0] | 295.0 [196.0 to 1157.0]

ADVERSE EVENTS:
Time Frame: 4 years, 6 months
Arm/Group | Active Comparator: Purified Isoflavones | Placebo Comparator: Methyl Cellulose Blend
Serious Adverse Events (participants affected / at risk) | 0/36 | 2/35
Other Adverse Events (participants affected / at risk) | 27/36 | 24/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Purified Isoflavones (N=36) | Placebo Comparator: Methyl Cellulose Blend (N=35)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Inoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Purified Isoflavones (N=36) | Placebo Comparator: Methyl Cellulose Blend (N=35)
Stomach cramps (Gastrointestinal disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Occasional Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, Belching (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, GI symptoms (Gastrointestinal disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Investigations - Other, Elevated total testosterone (Investigations) | 0 | 1
Investigations - Other, Low hemoglobin (Investigations) | 0 | 1
Investigations - Other, Low RBC (Investigations) | 0 | 2
Metabolism and nutrition disorders - Other, Low carbon dioxide (Metabolism and nutrition disorders) | 5 | 4
Metabolism and nutrition disorders - Other, Low globulin (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other, Low protein (Metabolism and nutrition disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Renal and urinary disorders - Other, Urination discomfort (Renal and urinary disorders) | 0 | 1
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastrointestinal disorder - Other, Tender stomach (Gastrointestinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Gastrointestinal disorder - Other, Darkening of stool (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, Soft stool (Gastrointestinal disorders) | 1 | 0
General disorders - Other, Feeling of fullness (General disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Investigations - Other, Elevated estradiol (Investigations) | 1 | 0
Investigations - Other, Low serum Co2 (Investigations) | 1 | 0
Investigations - Other, Low total testosterone (Investigations) | 1 | 0
Metabolism and nutrition disorders - Other, Elevated albumin (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, Low creatinine (Metabolism and nutrition disorders) | 2 | 0
Renal and urinary disorders - Other, Slow stream (Renal and urinary disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders, Other - Frequent urination (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders, Other - Frequent urination (night) (Renal and urinary disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0

LIMITATIONS AND CAVEATS:
Since the accrual of African American Men (AAM) was far lower than expected, this study was ultimately underpowered to detect small changes in specific biomarkers of disease progression proposed in men with localized prostate cancer (PCa).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes